CLINICAL TRIAL: NCT01833390
Title: Study of Hyperpolarized Xenon (MagniXene) in Patients With Obstructive Pulmonary Diseases (Asthma and COPD) to Assess Regional Lung Function by Delineating Regions of Abnormal Lung Ventilation
Brief Title: MagniXene MRI Use in Patients With Asthma and COPD to Assess Regional Lung Function by Delineating Ventilation Defects
Acronym: HXe-VENT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Xemed LLC (Industry)
Collaborators: University of Virginia (Other); National Institutes of Health (NIH) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MagniXene-087550-01; R44HL087550 (NIH)
Record Dates: First submitted 2013-04-01; First posted 2013-04-16 (Estimated); Last update posted 2015-03-11 (Estimated); Status verified 2015-02

CONDITIONS: Asthma; COPD; Healthy
Keywords: Hyperpolarized Xenon; HXe; MagniXene
MeSH Terms: conditions — Asthma; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- HXe MRI lung ventilation (Experimental): Each subject will inhale a dose of HXe gas (up to one liter HXe) while lying inside an MRI scanner. A high-resolution 3D map of the lung spaces filled with HXe gas will be acquired during a short breath-hold. Additionally, proton MRI of the chest cavity will be recorded during the same breath-hold for registering the lung boundaries. All subjects will undergo Pulmonary Function Tests. Subjects suffering from obstructive lung disease will have Tc-99m DTPA lung scintigraphy performed for comparing with HXe images.
  Interventions: Drug: HXe MRI lung ventilation

INTERVENTIONS:
Drug: HXe MRI lung ventilation — MagniXene (HXe) is an Investigational New Drug made of xenon noble gas. Through a physical process using alkali vapors and powerful lasers, xenon atoms have their nuclear spin preferentially aligned (hyperpolarized), thus offering a highly enhanced signal inside an MRI scanner. High-resolution images of the lung spaces are acquired within a short breath-hold after inhalation of HXe.
  Other Names: Hyperpolarized Xenon; MagniXene; HXe

SUMMARY:
The purpose of this clinical trial is to demonstrate hyperpolarized xenon (HXe) as a medical imaging drug (agent) for Magnetic Resonance Imaging (MRI) of the human lung ventilation.

DETAILED DESCRIPTION:
HXe MRI provides a diversity of imaging techniques for interrogating pulmonary function and lung microstructure. The most mature of these techniques utilizes HXe spin-density MRI to depict regional lung ventilation. Prior work suggests that ventilation imaging has utility in all obstructive lung diseases. This is a Phase II clinical trial to assess HXe MRI capability of providing qualitative and quantitative clinical information regarding lung ventilation. Proton and xenon images will be acquired within single breath holds on 28 subjects per year, including healthy volunteers and patients with COPD and asthma. All studies will include repeat scans and Pulmonary Function Tests (PFT). Ventilation scans with Technetium-99m (Tc-99m) diethylene-triamine-pentaacetate (DTPA) aerosol scintigraphy will be acquired on lung patients.

The primary goal of this aim is to validate the effectiveness of HXe ventilation MRI for delineating regions of normal and abnormal lung ventilation. To validate the regional depiction of ventilation, HXe MRI ventilation will be compared with nuclear medicine Tc-99m DTPA ventilation scintigraphy. The comparatively low spatial and temporal resolution of ventilation scintigraphy will limit this study to demonstrating only that HXe MRI ventilation is not inferior to the current clinical standard. Additionally, the concordance between measurements of the whole lung volume from both proton MRI and HXe MRI with PFT, the current clinical standard for lung volume measurement, will be assessed as a secondary outcome of the study.

ELIGIBILITY:
Inclusion Criteria (healthy subjects):

* Currently feeling well without respiratory symptoms.
* No history of lung disease.
* Never personally smoked (defined as less 100 cigarettes in their lifetime).

Inclusion Criteria (COPD subjects):

* Forced Expiratory Volume in 1 second (FEV1)<80% predicted OR FEV1 to Forced Vital Capacity (FVC) ratio <70%
* Smoking history >10 pack years
* Subjects should be at their clinical baseline on the day of imaging
* Subjects must be clinically stable in order to participate in the study

Inclusion Criteria (asthma subjects):

* Greater than 10% increase in FEV1 30-50 minutes after administration of albuterol;
* Subjects should be at their clinical baseline on the day of imaging;
* Subjects must be clinically stable in order to participate in the study.

Exclusion Criteria:

* Baseline oxygen requirement.
* Blood oxygen saturation of 92% less than as measured by pulse oximetry on the day of imaging.
* FEV1 percent predicted less than 25%.
* Pregnancy or lactation.
* Claustrophobia, inner ear implants, aneurysm or other surgical clips, metal foreign bodies in eye, pacemaker or other contraindication to MR scanning. Subjects with any implanted device that cannot be verified as MRI compliant will be excluded.
* Chest circumference greater than that of the xenon MR coil.
* History of congenital cardiac disease, chronic renal failure, or cirrhosis.
* Inability to understand simple instructions or to hold still for approximately 10 seconds.
* History of respiratory infection within 2 weeks prior to the MR scan.
* History of heart attack, stroke and/or poorly controlled hypertension.
* Known hypersensitivity to albuterol or any of its components, or levalbuterol.

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2011-09; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
HXe MRI delineation of regions with abnormal lung ventilation in asthma and COPD patients | three years
  Depiction of ventilation defects with HXe MRI is not worse than presently accepted clinical method, Tc-99m DTPA scintigraphy, as judged by skilled readers and software analysis. The primary outcome variable will be binary: if ventilation is detected the value is 1, the value is 0 otherwise (defect). The level of agreement between HXe MRI and Tc-99m DTPA will be statistically calculated.

SECONDARY OUTCOMES:
Ventilated volume of the lungs determined by HXe MRI | three years
  A secondary outcome will be HXe MRI capability of describing parameters of the lung physiology, such as the ventilated volume of the lungs as compared to that extracted from imaging the pleural cavity via proton MRI for healthy subjects and from the pulmonary function tests for lung disease patients.
Number of ventilation defects in COPD and asthma patients | three years
  The agreement between the number of ventilation defects as determined by skilled readers from HXe MRI and Tc-99m DTPA scintigraphy will be studied based on an extension of the Bland Altman statistical method for repeated measures data.

CONTACTS AND LOCATIONS:
Overall Officials: Talissa A Altes, M.D., Principal Investigator — University of Virginia; Iulian C Ruset, PhD, Principal Investigator — Xemed LLC
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States